CLINICAL TRIAL: NCT02061969
Title: A Randomized Controlled Study Comparing a DPP4 Inhibitor (Linagliptin) and Basal Insulin (Glargine) in Long-Term Care Residents With Type 2 Diabetes
Brief Title: ADA Linagliptin in Long Term Care
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Emory University (Other)
Collaborators: American Diabetes Association (Other)
Responsible Party: Principal Investigator, Guillermo Umpierrez, MD, Professor of Medicine, Emory University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IRB00071545; IRB00071946 (Other: VA site IRB number)
Record Dates: First submitted 2014-02-11; First posted 2014-02-13 (Estimated); Results first posted 2018-08-22 (Actual); Last update posted 2018-08-22 (Actual); Status verified 2018-07

CONDITIONS: Diabetes
Keywords: nursing home facility; long-term care facility; older patients; elderly patients; hyperglycemia; type 2 diabetes
MeSH Terms: conditions — Diabetes Mellitus; Hyperglycemia; Diabetes Mellitus, Type 2 | interventions — Linagliptin; Insulin Glargine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Insulin glargine (Active Comparator): Insulin glargine starting at 0.1 unit/kg/day added to ongoing metformin if the patient is already on it. The duration will be for a 6-month period.
  Interventions: Drug: insulin glargine
- linagliptin (Experimental): Oral linagliptin 5mg once daily added to ongoing metformin if the patient is already on it. The duration will be for a 6-month period.
  Interventions: Drug: linagliptin

INTERVENTIONS:
Drug: linagliptin — 5mg linagliptin tablets
  Other Names: Tradjenta
  Arms: linagliptin
Drug: insulin glargine
  Other Names: Lantus
  Arms: Insulin glargine

SUMMARY:
This is a study to determine whether glycemic control, as measured by change in HbA1c and frequency of hypoglycemia, is different between treatment with linagliptin (Tradjenta®) and basal insulin in long term care residents(LTC) with Type 2 diabetes(T2D). Patients with poorly controlled diabetes (HbA1c >7.5%) will be randomized to a 6-month intervention with linagliptin or glargine insulin (± metformin for both treatments). Our hypothesis is that treatment with linagliptin, a once daily DPP4-inhibitor, will result in similar improvement in glucose control but in a lower rate of hypoglycemia than insulin treatment in LTC residents with T2D. We will also determine differences in clinical outcome, resource utilization, and hospitalization costs between LTC residents with T2D treated with linagliptin and basal and correction insulin. We will compare differences in complications (infectious and non-infectious, neurological and cardiovascular events), emergency room visits and hospitalizations between groups during the 6 months of intervention.

ELIGIBILITY:
Inclusion Criteria:

1. Males or females with known history of type 2 diabetes, treated with diet, OADs as monotherapy or in combination therapy (excluding DPP4 inhibitors), or sliding scale insulin.
2. Subjects with HbA1c > 7.5% and/or any blood glucose greater than or equal to 180 mg/dL

Exclusion Criteria:

1. Subjects with a history of type 1 diabetes or with a history of diabetic ketoacidosis
2. Treatment with insulin or GLP1 analogs during the past 3 months prior to admission.
3. Recurrent severe hypoglycemia or hypoglycemic unawareness.
4. Subjects with history of gastrointestinal obstruction or gastroparesis.
5. Patients with acute or chronic pancreatitis or pancreatic cancer.
6. Patients with clinically significant hepatic disease (cirrhosis, jaundice, end-stage liver disease, portal hypertension) and elevated ALT and AST > 3 times upper limit of normal, or significantly impaired renal function (GFR < 45 ml/min).
7. Treatment with corticosteroids, parenteral nutrition and immunosuppressive treatment.
8. Mental condition rendering the subject unable to understand the nature and scope of the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 140 (Actual)
Dates: Start 2014-04-25; Primary Completion 2017-04-10 (Actual); Study Completion 2017-04-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Guillermo Umpierrez, MD, Principal Investigator — Emory University
Locations (4):
- United States (4):
  - Crestvew Nursing Home, Atlanta, Georgia
  - Budd Terrace Nursing Home, Atlanta, Georgia
  - Wesley Woods Nursing Home, Atlanta, Georgia
  - VA Nursing Home, Decatur, Georgia

REFERENCES:
- [Derived] Umpierrez GE, Cardona S, Chachkhiani D, Fayfman M, Saiyed S, Wang H, Vellanki P, Haw JS, Olson DE, Pasquel FJ, Johnson TM 2nd. A Randomized Controlled Study Comparing a DPP4 Inhibitor (Linagliptin) and Basal Insulin (Glargine) in Patients With Type 2 Diabetes in Long-term Care and Skilled Nursing Facilities: Linagliptin-LTC Trial. J Am Med Dir Assoc. 2018 May;19(5):399-404.e3. doi: 10.1016/j.jamda.2017.11.002. Epub 2017 Dec 27. PMID 29289540

RESULTS

PARTICIPANT FLOW:
Groups:
- Insulin Glargine: Insulin glargine starting at 0.1 unit/kg/day added to ongoing metformin if the patient is already on it. The duration will be for a 6-month period.
  Insulin glargine
Period: Overall Study
Arm/Group | Insulin Glargine | Linagliptin
Started | 73 | 67
Completed | 73 | 67
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Insulin Glargine | Linagliptin | Total
Number analyzed (Participants) | 73 | 67 | 140
Age, Continuous [Mean (Standard Deviation); unit: years] | 71.5 (13) | 68 (14) | 69.8 (13)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 48 | 35 | 83
  Male | 25 | 32 | 57
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 42 | 42 | 84
  White | 30 | 22 | 52
  More than one race | 1 | 3 | 4
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 73 | 67 | 140

OUTCOME MEASURES:

1. Primary Outcome: Mean Fasting Blood Glucose Level
Description: The primary endpoint of the study is differences between treatment groups in mean fasting blood glucose level in LTC residents with poorly controlled diabetes.
Time Frame: 6 months
Measure: Mean (Standard Deviation); unit: mg/dl
Arm/Group | Insulin Glargine | Linagliptin
Number analyzed (Participants) | 73 | 67
mg/dl | 136.4 (35) | 131.2 (27)

2. Secondary Outcome: HbA1c
Description: HbA1c at 6 month
Time Frame: 6 months
Measure: Mean (Standard Deviation); unit: percent of glycosylated hemoglobin
Arm/Group | Insulin Glargine | Linagliptin
Number analyzed (Participants) | 73 | 67
percent of glycosylated hemoglobin | 6.58 (0.7) | 6.82 (0.6)

3. Secondary Outcome: Number of Hypoglycemic Events < 70mg/dl
Description: total number of hypoglycemic events (<70 mg/dl)
Time Frame: over 6 months
Measure: Number; unit: events
Arm/Group | Insulin Glargine | Linagliptin
Number analyzed (Participants) | 73 | 67
events | 136 | 3

4. Secondary Outcome: Number of Hypoglycemic Events < 40mg/dl
Description: total number of severe hypoglycemia (< 40 mg/dl).
Time Frame: over 6 months
Measure: Number; unit: events
Arm/Group | Insulin Glargine | Linagliptin
Number analyzed (Participants) | 73 | 67
events | 3 | 0

5. Secondary Outcome: Total Daily Dose of Insulin
Description: Total daily dose of insulin (units)
Time Frame: over 6 months
Measure: Mean (Standard Deviation); unit: U/day
Arm/Group | Insulin Glargine | Linagliptin
Number analyzed (Participants) | 73 | 67
U/day | 12.0 (9.9) | 4.03 (1.7)

6. Secondary Outcome: Changes in Cognitive Function
Description: Data on changes in cognitive function were not collected
Time Frame: over 6 months
Population: Data were not collected
Arm/Group | Insulin Glargine | Linagliptin
Number analyzed (Participants) | 0 | 0

7. Secondary Outcome: Number of Participants With Acute Complications
Description: Number of Participants with Acute Complications (urinary tract infections, pneumonia, bedsores, diabetic foot infection).
Time Frame: over 6 months
Measure: Count of Participants; unit: Participants
Arm/Group | Insulin Glargine | Linagliptin
Number analyzed (Participants) | 73 | 67
Participants | 8 | 5

8. Secondary Outcome: Total Number of Emergency Room Visits
Description: Total number of emergency room visits during the study period
Time Frame: 6 months
Measure: Number; unit: visits
Arm/Group | Insulin Glargine | Linagliptin
Number analyzed (Participants) | 73 | 67
visits | 3 | 0

9. Secondary Outcome: Total Number of Hospital Visits
Description: Total number of hospital visits during the study period
Time Frame: 6 months
Measure: Number; unit: visits
Arm/Group | Insulin Glargine | Linagliptin
Number analyzed (Participants) | 73 | 67
visits | 6 | 7

10. Secondary Outcome: Total Number of Complications
Description: Total number of complications including urinary tract infections, pneumonia, diabetic foot infection, cardiac complications including myocardial infarction and heart failure, cerebrovascular accidents, and acute kidney injury and mortality.
Time Frame: 6 months
Measure: Number; unit: events
Arm/Group | Insulin Glargine | Linagliptin
Number analyzed (Participants) | 73 | 67
events | 22 | 16

11. Secondary Outcome: Incidence of Acute Kidney Injury
Description: Acute kidney injury in LTC Residents Treated with Basal Insulin and Linagliptin Therapy
Time Frame: over 6 months
Measure: Number; unit: events
Arm/Group | Insulin Glargine | Linagliptin
Number analyzed (Participants) | 73 | 67
events | 2 | 1

12. Secondary Outcome: Mortality
Description: Mortality is defined as death occurring during admission at the LTC facility
Time Frame: over 6 months
Measure: Count of Participants; unit: Participants
Arm/Group | Insulin Glargine | Linagliptin
Number analyzed (Participants) | 73 | 67
Participants | 0 | 2

ADVERSE EVENTS:
Time Frame: 6 months
Arm/Group | Insulin Glargine | Linagliptin
All-Cause Mortality (participants affected / at risk) | 0/73 | 2/67
Serious Adverse Events (participants affected / at risk) | 6/73 | 4/67
Other Adverse Events (participants affected / at risk) | 16/73 | 12/67
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Insulin Glargine (N=73) | Linagliptin (N=67)
Hospitalized for Altered Mental Status (Psychiatric disorders) | 0 (0) | 1 (1)
Hospitalized for repair craninectomy (Surgical and medical procedures) | 1 (1) | 0 (0)
Hospitalized for aspiration pneumonia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Hospitalization for pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Hospitalization for congestive heart failure ( exacerbation (Cardiac disorders) | 1 (1) | 0 (0)
Right stump infection (Infections and infestations) | 1 (1) | 0 (0)
Hospitalized for brain edema (Nervous system disorders) | 1 (1) | 0 (0)
Hospitalized for severe aortic stenosis (Cardiac disorders) | 0 (0) | 1 (1)
Amputation of the left 2nd toe (Surgical and medical procedures) | 0 (0) | 1 (1)
Wound infection (Infections and infestations) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Insulin Glargine (N=73) | Linagliptin (N=67)
Chest pain (Cardiac disorders) | 0 (0) | 1 (1)
Shingels (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2)
Hematuria (Renal and urinary disorders) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 0 (0) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 0 (0) | 1 (1)
Urinary Tract Infection (Renal and urinary disorders) | 6 (6) | 3 (3)
Pneumonia (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1)
Acute Kidney Injury (Renal and urinary disorders) | 0 (0) | 1 (1)
Acute renal failure (Renal and urinary disorders) | 3 (3) | 0 (0)
Bradicardia (Cardiac disorders) | 1 (1) | 0 (0)
Hypotension (Cardiac disorders) | 1 (1) | 0 (0)
Anemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Penile infection (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Fall (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-08-11): https://cdn.clinicaltrials.gov/large-docs/69/NCT02061969/Prot_SAP_000.pdf